CLINICAL TRIAL: NCT04303286
Title: The Effect of Gut Microbiota on Postoperative Liver Function Recovery in Patients With Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Zhang Bi Xiang, MD, Chairman of Department of General Surgery, Tongji Hospital
Other Study IDs: TJ-IRB20191223
Record Dates: First submitted 2020-03-05; First posted 2020-03-11 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Gut Microbiota; Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — feces, whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Recovery Group: The liver function of HCC patients on the fifth day after the operation is recovered.
- Recovery Delay Group: The liver function of HCC patients on the fifth day after the operation is delayed recovered.
- Control Group: The patients on benign disease of the liver

SUMMARY:
The purpose of this study was to explore the correlation between postoperative recovery of liver function and gut microbiota in patients with hepatocellular carcinoma (HCC). Liver resection patients were divided into the recovery group and the recovery delay group according to the recovery level of liver function on the fifth day after the operation. Benign liver disease was used as a control. Statistical analysis was performed to compare the differences in gut microbiota between the three groups. Then, fecal microbiota transplantation was performed in a mouse hepatectomy model. Through this study, the investigators hope to understand the relationship between gut microbiota and postoperative recovery of liver function in patients with hepatocellular carcinoma, so as to provide a new therapeutic direction for patients in the aspect of perioperative liver function recovery.

DETAILED DESCRIPTION:
Primary hepatocellular carcinoma (HCC) is one of the most common malignant tumors in the world. At present, surgery is the first choice and the most effective way to treat it. Based on the case review, the investigators found that the recovery rate of perioperative liver function was correlated with survival. Therefore, it is of great clinical significance to improve the recovery rate of postoperative liver function. Gut microbiota participate in many physiological activities of human body, such as metabolic regulation, immune homeostasis and hormone regulation. However, gut microbiota imbalance, excessive growth of pathogenic microorganisms and changes in intestinal mucosal permeability lead to intestinal bacterial ectopia and bacterial metabolites entering the liver through enterohepatic circulation. The continuous inflammatory stimulation aggravate the progress of liver disease. Therefore, it is helpful to explore the influence of gut microbiota on postoperative liver function recovery and find out the different microbiota, in order to improve the postoperative liver function recovery rate, shorten the perioperative hospital stay and prolong the survival of patients.

According to the recovery level of liver function on the fifth day after the operation, liver resection patients on HCC were divided into the recovery group and the recovery delay group which comparing on the time point of before the surgery and five days after the surgery. The patients on benign liver disease were used as a control. The investigators attempt to identify the differential microbiota and validate this finding in a mouse hepatectomy model.

ELIGIBILITY:
Inclusion Criteria:

* The patient is diagnosed with liver cancer by b-mode ultrasonography before the surgery.
* There is no antibiotic treatment, no severe diarrhea and regular diet within two weeks before the surgery.
* It perform laparoscopic or open hepatectomy.
* The postoperative pathological diagnosis is hepatocellular carcinoma.

Exclusion Criteria:

* No hepatectomy is performed during the operation.
* The patient is't hepatocellular carcinoma due to the postoperative pathological diagnosis.
* No stool samples are collected during the perioperative period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort are the patients from the hepatic surgery of Tongji hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Diversity analysis | Before the surgery
  We will use 16S rRNA sequencing to measure fecal sample. The alpha and beta diversity of gut microbiota between the groups will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity.
Diversity analysis | Five days after the surgery
  We will use 16S rRNA sequencing to measure fecal sample. The alpha and beta diversity of gut microbiota between the groups will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity.
Species composition analysis | Before the surgery
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the community histogram, the community heatmap and the Wayne map will be used to analyze the species composition of the sample, in order to explore the relationship between the species and the sample, and analyze the key microflora in the sample.
Species composition analysis | Five days after the surgery
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the community histogram, the community heatmap and the Wayne map will be used to analyze the species composition of the sample, in order to explore the relationship between the species and the sample, and analyze the key microflora in the sample.
Species differential analysis | Before the surgery
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the PCA、PCoA and NMDS analysis will be used to assess the similarities and differences in species composition between groups. To further screen the species with significant differences, the LEfSe difference discriminant analysis will be used.
Species differential analysis | Five days after the surgery
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the PCA、PCoA and NMDS analysis will be used to assess the similarities and differences in species composition between groups. To further screen the species with significant differences, the LEfSe difference discriminant analysis will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Bixiang Zhang, Study Chair — Tongji Hospital; Jingjing Yu, Principal Investigator — Tongji Hospital
Locations (1):
- The hepatic surgery of Tongji hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Yu J, Zhu P, Shi L, Gao N, Li Y, Shu C, Xu Y, Yu Y, He J, Guo D, Zhang X, Wang X, Shao S, Dong W, Wang Y, Zhang W, Zhang W, Chen WH, Chen X, Liu Z, Yang X, Zhang B. Bifidobacterium longum promotes postoperative liver function recovery in patients with hepatocellular carcinoma. Cell Host Microbe. 2024 Jan 10;32(1):131-144.e6. doi: 10.1016/j.chom.2023.11.011. Epub 2023 Dec 12. PMID 38091982